CLINICAL TRIAL: NCT01560897
Title: Investigating Project of the Functional C13 Test
Brief Title: Investigating Project of the Functional C13 Test "Pilot Study"
Acronym: PIL001
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pilot Study
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Disorder of the Urea Cycle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C13 (Experimental): The dose of sodium [1-13C] acetate is calculated according to patient weight (27mg/kg) or (0.33 mmol / kg).
  Interventions: Drug: Oral C13

INTERVENTIONS:
Drug: Oral C13 — Ingestion of C13 and follow up of the ureogenesis

SUMMARY:
The aim of this pilot study is to evaluate the validity and reproducibility of a functional test "Test C13" ureogenesis to measure in vivo, using the methodology Laboratory of Metabolic Diseases of "Cliniques Universitaires Saint-Luc"

ELIGIBILITY:
Inclusion Criteria:

* healthy or with a disorder of the urea cycle

Exclusion Criteria:

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Subject with a disorder of the urea cycle | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Saint Luc, Brussels, Belgium